CLINICAL TRIAL: NCT04149327
Title: Systemic Antibiotic Therapy (Amoxicillin Plus Metronidazole) as an Adjunct to Initial Non-surgical Treatment of Peri-implantitis; a Single Blind Randomized Controlled Study
Brief Title: Systemic Amoxicillin Plus Metronidazole in Peri-implantitis Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL41441.042.12
Record Dates: First submitted 2019-10-26; First posted 2019-11-04 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Peri-implantitis; Periodontal Diseases
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotics group (Experimental): Patients will receive full-mouth mechanical cleansing of both implants and remaining dentition using ultrasonic instruments (EMS®) and hand instruments (scalers and curettes) in one or multiple sessions (max. 4). Prior to each session patients will rinse their mouth using 0.12% chlorhexidine + 0.05% cetylpyridinium chloride without alcohol during 30 seconds. At the final session all previously cleaned areas will be re-examined and cleaned. At the end of the final treatment session, the dental hygienist will give the patients an envelop containing a recipe for medication consisting of 500 mg amoxicillin and 500 mg metronidazole to be taken every 8 hours for the following 7 days plus a recipe for 500 ml mouthrinse (0.12% chlorhexidine + 0.05% cetylpyridinium chloride without alcohol, Perio-Aid®). After the final session patients will rinse their mouth using that mouthrinse twice daily during 30 seconds for 2 weeks.
  Interventions: Drug: amoxicillin 500 mg + metronidazole 500 mg; Procedure: non-surgical periodontal and peri-implant treatment
- Control group (Active Comparator): Patients will receive full-mouth mechanical cleansing of both implants and remaining dentition using ultrasonic instruments (EMS®) and hand instruments (scalers and curettes) in one or multiple sessions (max. 4). Prior to each session patients will rinse their mouth using 0.12% chlorhexidine + 0.05% cetylpyridinium chloride without alcohol during 30 seconds. At the final session all previously cleaned areas will be re-examined and cleaned. At the end of the final treatment session, the dental hygienist will give the patients an envelop containing a recipe for 500 ml mouthrinse (0.12% chlorhexidine + 0.05% cetylpyridinium chloride without alcohol, Perio-Aid®). After the final session patients will rinse their mouth using that mouthrinse twice daily during 30 seconds for 2 weeks.
  Interventions: Procedure: non-surgical periodontal and peri-implant treatment

INTERVENTIONS:
Drug: amoxicillin 500 mg + metronidazole 500 mg — 500 mg amoxicillin and 500 mg metronidazole to be taken every 8 hours for 7 days
  Arms: Antibiotics group
Procedure: non-surgical periodontal and peri-implant treatment — Patients are instructed on how to perform proper oral hygiene measures using an electric toothbrush, interdental brushes (to be used in combination with Corsodyl® gel) and floss (Oral-B® superfloss or Meridol® floss, at implants only).
  Patients will receive full-mouth mechanical cleansing of both implants and remaining dentition using ultrasonic instruments (EMS®) and hand instruments (scalers and curettes) in one or multiple sessions (max. 4). Prior to each session patients will rinse their mouth using 0.12% chlorhexidine + 0.05% cetylpyridinium chloride without alcohol during 30 seconds. At the final session all previously cleaned areas will be re-examined and cleaned.

SUMMARY:
The primary objective of this controlled clinical trial is to evaluate the clinical effect of systemic amoxicillin plus metronidazole therapy in conjunction with initial non-surgical treatment of peri-implantitis. The secondary objective is to assess the microbiological effectiveness of this peri-implantitis treatment approach.

The present study is a single-blind, randomized controlled clinical trial. Adult patients with at least one endosseous implant in the oral cavity with clinical and radiographical evidence of periimplantitis will be included in this study.

Patients with implants affected by peri-implantitis will receive initial periodontal treatment existing of oral hygiene instructions and mechanical cleansing of both implants and remaining dentition. Immediately after initial periodontal therapy patients will be instructed to rinse their mouth with 0.12% chlorhexidine + 0.05% cetylpyridinium chloride without alcohol twice daily during 30 seconds for 2 weeks. Additionally patients will receive a recipe for medication consisting of 500 mg amoxicillin and 500 mg metronidazole to be taken every 8 hours for the following 7 days or no recipe.

The main study parameter is the mean peri-implant bleeding score.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years of age;
* The patient has at least one endosseous implant in the oral cavity with clinical and radiographical signs of peri-implantitis. Peri-implantitis is defined as a loss of marginal bone ≥ 2 mm as compared to the shoulder of the implant (the level at which the bone is normally located immediately after implant placement), in combination with bleeding and/or suppuration on probing and a peri-implant probing depth ≥ 5 mm;
* The implants have been in function for at least two years;
* The patient is capable of understanding and giving informed consent.

Exclusion Criteria:

* Medical and general contraindications for the surgical procedures;
* A history of local radiotherapy to the head and neck region;
* Pregnancy and lactation;
* Uncontrolled diabetes (HbA1c < 7% or < 53 mmol/mol)
* Mononucleosis infectiosa
* Organic neurological disorders
* Use of antibiotics during the last 3 months;
* Known allergy to amoxicillin, metronidazole or chlorhexidine;
* Long-term use of anti-inflammatory drugs;
* Full edentulism (no remaining teeth, only implants)
* Incapability of performing basal oral hygiene measures as a result of physical or mental disorders;
* Implants placed in areas augmented with autogenous bone from the crista iliac region;
* Implants placed in skin grafted areas;
* Implants with bone loss exceeding 2/3 of the length of the implant or implants with bone loss beyond the transverse openings in hollow implants;
* Implant mobility;
* Implants at which no position can be identified where proper probing measurements can be performed;
* Previous surgical treatment of the peri-implantitis lesions;
* Previous non-surgical treatment of the peri-implantitis lesions during the last 6 months (scaling or curettage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
change from baseline mean peri-implant bleeding score at 3 months | 3 months after therapy
  in percentages ranging from 0 (no change) to 100 (improvement)

SECONDARY OUTCOMES:
change from baseline full-mouth periodontal bleeding score at 3 months | 3 months after therapy
  in percentages ranging from 0 (no change) to 100 (improvement)
change from baseline mean peri-implant and baseline full-mouth periodontal suppuration on probing score at 3 months | 3 months after therapy
  in percentages ranging from 0 (no change) to 100 (improvement)
change from baseline mean peri-implant and full-mouth periodontal probing pocket depth at 3 months | 3 months after therapy
  in millimeters ranging from 0 (no change) to high (improvement)
change from baseline mean peri-implant and full-mouth periodontal plaque score at 3 months | 3 months after therapy
  in percentages ranging from 0 (no change) to 100 (improvement)
change from baseline marginal soft tissue level at 3 months | 3 months after therapy
  in millimeters ranging from 0 (no change) to high (worsening)
change from baseline radiographic marginal peri-implant bone level at 3 months | 3 months after therapy
  in millimeters ranging from 0 (no change) to high (worsening)
change from baseline in detection frequency of 7 periodontal pathogens potentially residing in the peri-implant and periodontal area at 3 months | 3 months after therapy
number of patients in need for additional surgery at teeth and implants | 3 months after therapy
number of patients with implant failure, defined as implant mobility of previously clinically osseointegrated implants and removal of non-mobile implants because of progressive marginal bone loss or infection | 3 months after therapy
number of patients with tooth loss, defined as removal of teeth because of progressive marginal bone loss or infection | 3 months after therapy
number of patients with adverse events related to the treatment | 3 months after therapy